CLINICAL TRIAL: NCT02368964
Title: Treatment for Final Follicular Maturation Induction in Patients With Previous High Ratio of Immature Oocytes
Brief Title: IVF Treatment in Women With Immature Oocytes in Previous Cycle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Aya Mohr-Sasson, Doctor, Sheba Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHEBA-14-1817-YH-CTIL
Record Dates: First submitted 2015-02-10; First posted 2015-02-23 (Estimated); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Infertility
Keywords: double triggering; Oocyte maturation; GNRH Agonist; hCG; IVF treatment; immature oocytes
MeSH Terms: conditions — Infertility | interventions — Gonadotropin-Releasing Hormone; Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose hCG (Experimental): The hCG group- will be triggered for final follicular maturation with high dose hCG (500 mcg)-38 hours prior to oocyte aspiration
  Interventions: Drug: high dose hCG 500 mcg
- Double trigger (Experimental): Double trigger Group- will receive GnRH agonist (Decapeptyl 0.2mg) 40 hours prior to oocyte aspiration and hCG (250mcg) 34 hours prior to the oocyte aspiration
  Interventions: Drug: GnRH agonist 0.2 mg + hCG 250 mcg

INTERVENTIONS:
Drug: GnRH agonist 0.2 mg + hCG 250 mcg — Treatment for triggering
  Other Names: GnRH agonist - Decapeptyl , hCG - Ovitrelle
  Arms: Double trigger
Drug: high dose hCG 500 mcg — Treatment for triggering
  Other Names: Ovitrelle
  Arms: High dose hCG

SUMMARY:
In standard IVF stimulation cycle,human chorionic gonadotropin (hCG) is usually used at the end of controlled ovarian hyperstimulation (COH) as a surrogate to only the luteinizing hormone (LH) surge. Yet, the last dose of follicle stimulating hormone (FSH) is usually given between 12-24 hours before the hCG triggering dose.One protocol used at the investigators unit, after a cycle with low proportion of mature oocytes per number oocytes retrieved, is triggering with high dose hCG (500 mcg)-38 hours prior to oocyte aspiration.

Lately, new researches showed that dual triggering of final oocyte maturation with a combination of GnRH- agonist and hCG, could improve the live-birth rate of normal responders undergoing the GnRH-antagonist COH protocol

Another treatment option is high dose hCG. Only few case reports have described the use of high dose hCG after aspiration of non mature oocytes at a previous cycle. At the investigators IVF unit, patients with previous history of high percentage of immature oocytes retrieved, are triggered at the following cycle, either with double trigger or with high dose of hCG decided by the physician consulting the patient. It is still not known with which way of triggering more mature oocytes is retrieved.

The aim of this study is to perform a prospective randomized controlled study in patients with low proportion of mature-MII oocytes oocytes (<75%) per number oocytes retrieved, despite normal response to controlled ovarian hyperstimulation ( COH ) comparing cycles triggered with high dose hCG to those triggered with hCG+GnRH agonist.

DETAILED DESCRIPTION:
Patients will be prospectively randomized into two groups. The randomization will be organized through the computer. The hCG group- will be triggered for final follicular maturation with high dose hCG (500 mcg)-38 hours prior to oocyte aspiration, and the Double trigger Group- will receive gonadotropin-releasing hormone (GnRH) agonist (Decapeptyl 0.2mg) 40 hours prior to oocyte aspiration and hCG (250mcg) 34 hours prior to the oocyte aspiration. All patients will be supplemented with the same progesterone preparation( Crinone gel 8% once a day) for luteal support. Women that suffer from vaginal spotting or vaginal bleeding during the luteal phase will receive supplementation of Geston 50MG intramuscular once every 2 days.

At the day of oocyte aspiration, blood will be drawn for serum LH, FSH, estrogen (E2) and progesterone. Moreover, clear follicular fluid will be collected and tested for LH, FSH, E2 and progesterone levels.

ELIGIBILITY:
Inclusion Criteria:

* Patients with low proportion of mature-MII oocytes oocytes (75%) per number oocytes retrieved at the prior IVF cycle
* Age between 18-42

Exclusion Criteria:

* Women with high ovarian response:anti-mullerian hormone ( AMH) >5, antral follicle count ( AFC) >15
* more than 20 oocytes retrieved at the prior cycle.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Number MII oocytes per number of oocytes retrieved | day of retrieving the oocytes
  Rate of mature oocytes from total oocytes retrieved

SECONDARY OUTCOMES:
Total oocytes | day of retrieving the oocytes
Pregnancy rate | Two weeks from induction of ovulation
Number of top quality embryos | day of retrieving the oocytes

CONTACTS AND LOCATIONS:
Overall Officials: Aya Mohr Sasson, M.D, Principal Investigator — Sheba Medical Center - IVF Unit
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel

REFERENCES:
- [Background] Lamb JD, Shen S, McCulloch C, Jalalian L, Cedars MI, Rosen MP. Follicle-stimulating hormone administered at the time of human chorionic gonadotropin trigger improves oocyte developmental competence in in vitro fertilization cycles: a randomized, double-blind, placebo-controlled trial. Fertil Steril. 2011 Apr;95(5):1655-60. doi: 10.1016/j.fertnstert.2011.01.019. PMID 21315341
- [Background] Lin MH, Wu FS, Lee RK, Li SH, Lin SY, Hwu YM. Dual trigger with combination of gonadotropin-releasing hormone agonist and human chorionic gonadotropin significantly improves the live-birth rate for normal responders in GnRH-antagonist cycles. Fertil Steril. 2013 Nov;100(5):1296-302. doi: 10.1016/j.fertnstert.2013.07.1976. Epub 2013 Aug 28. PMID 23993928
- [Background] Zilberberg E, Haas J, Dar S, Kedem A, Machtinger R, Orvieto R. Co-administration of GnRH-agonist and hCG, for final oocyte maturation (double trigger), in patients with low proportion of mature oocytes. Gynecol Endocrinol. 2015 Feb;31(2):145-7. doi: 10.3109/09513590.2014.978850. Epub 2014 Nov 11. PMID 25385007